CLINICAL TRIAL: NCT06759896
Title: Comparison Between Protraction Facemask and Upper Partial Fixed Appliance for Early Class III Intervention: a Randomized Controlled Trial
Brief Title: Comparison Between Protraction Facemask and Upper Braces for Underbite Correction in Growing Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Nur Farisya Binti Shamsuddin, Dr, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DF CD 2419/0055 (P)
Record Dates: First submitted 2024-12-20; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Anterior Crossbite; Class III Malocclusion in Growing Patients
Keywords: Randomized controlled trial; anterior crossbite

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial with 2 arm parallel
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 - Protraction facemask (Active Comparator): Patients assigned to Arm 1 will utilize the Petit protraction facemask, in conjunction with a rapid maxillary expansion (RME).
  Interventions: Device: Protraction facemask
- Arm 2 - Upper partial fixed appliance (Active Comparator): Patient allocated in Arm 2 will use upper partial fixed appliance / 2 by 4 appliance on their for upper incisors and molar band on upper 1st molars
  Interventions: Device: Upper partial fixed appliance

INTERVENTIONS:
Device: Protraction facemask — Patients assigned to intervention 1 will utilize the Petit protraction facemask, in conjunction with a rapid maxillary expansion (RME). This facemask consists of a forehead pad and chin pad linked by a sturdy steel support rod.
  Arms: Arm 1 - Protraction facemask
Device: Upper partial fixed appliance — Upper partial fixed appliance / 2 by 4 appliance will be used in this study by using bracket set (119-142 Unitek™ Gemini Bracket MBT™ U/L 5x5 0T-Cuspid 3Hk) with molar bands (3M™ Victory Series™ First Molar Bands) or buccal tubes (3M™ Victory Series™ Superior Fit Buccal Tubes) and upper nickel titanium archwires (3M™ Unitek™ Nitinol Heat-activated Archwire) and upper stainless steel archwires (3M™ Unitek™ Permachrome Standard Archwire) .
  Arms: Arm 2 - Upper partial fixed appliance

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of a protraction facemask and upper partial fixed appliance in correcting anterior crossbite in growing children with class III malocclusion. It will also learn about the patients perceptions of these treatments. The main questions it aims to answer are:

i. What is the rate of success in achieving anterior crossbite correction with the protraction facemask and upper partial fixed appliance? ii. Are there any significant differences in the dental, skeletal and soft tissue outcomes between the two treatment groups? iii. What are the patient's perceptions associated with each treatment modality received.

iv. What is the incidence of adverse effects or complications and breakages associated with each treatment modality?

Participants will be randomly assigned to one of two groups: 1) protraction facemask; or 2) upper partial fixed appliance. After investigators decide which group participants will be in, investigators will take some standard records for the study before starting the treatment. These records include:

1. Making moulds of their teeth to create study models
2. Taking a side-view X-ray of their head (called a lateral cephalometric radiograph)

Additionally, the participant will need to fill out a quick 5-minute survey called the Child Perceptions Questionnaire 8-10 (CPQ8-10). It has 25 short questions. The participant will do this survey at four different times: 1) before starting the treatment; 2) 3 months into the treatment; 3) 6 months into the treatment; and 4) after the treatment is done.

Investigators will set up appointments for the treatment based on the type assigned. Once the treatment starts, investigators will see the participant every six weeks until it is finished.

If the participant gets a protraction facemask, investigators will put a fixed expander appliance in the mouth at the palate. Investigators will teach them how to activate the appliance once a day for seven days. Afterwards, the participant will use the protraction facemask with elastics connecting the appliance in the mouth and the protraction facemask. The participant must wear it for 14 hours a day, at night.

If the participants gets an upper fixed partial appliance, investigators will bond upper fixed appliances in the mouth.

Investigators will teach the child how to clean the appliance and their mouth to avoid any potential problems or side effects during the treatment.

DETAILED DESCRIPTION:
1. Orthodontic assessment, consent and records taking All eligible patients identified at the Faculty of Dentistry, Universiti Malaya, will be scheduled for an orthodontic assessment during the research sessions. An explanation regarding the research objectives, interventions, randomization for treatment and details on protocols of each interventions will be given to the patient as written in the patient's information sheet. Patient will be reminded that they have to receive whatever treatment allocated to them with an open heart once they consented. Once patient agreed, further assessment will be done. If patient or parents not agree, their name will be put under waiting list for orthodontic treatment in this faculty. Following the extraoral and intraoral assessment, patient's parents or carer will have to sign a consent form. Then, study model impressions will be made using alginate Kromopan Type I Lascod, and bite registration will be done using modeling wax. Intraoral and extraoral photographs will be captured using a Canon EOS RP DSLR camera. Subsequently, appointments for dental panoramic tomography and lateral cephalometric radiography will be arranged at the X-ray Department, Faculty of Dentistry, Universiti Malaya.
2. Lateral cephalometric analysis In this study, Webceph Software Version 1.5.0 will be used for digital cephalometric analysis to assess skeletal and soft tissue of the patient. Soft copies of lateral cephalometric radiographs will be coded or named randomly by an individual assistant then uploaded to Webceph, and landmarks for skeletal and soft tissue analysis will be verified before conducting the analysis. All patients with ANB value equal to and less than 0 will be included in this study.
3. Interventions allocation All eligible patients will be randomized to determine their intervention as explained in 3.5.1. Further planning for their next appointment will be done as listed below

   1. Intervention 1 - Protraction facemask Overjet, overbite, canine and molar relationship will be measured from the study model and recorded in a data collection form. Then, appointment will be given for impression taking to construct the Rapid Maxillary Expansion (RME).
   2. Intervention 2 - Upper partial fixed appliance Overjet, overbite, canine and molar relationship will be measured from the study model and recorded in a data collection form. Then, an appointment for separators insertion will be arranged a week before appointment for the band and bond up procedures.
4. Treatment phase Before undergoing either intervention, all patients will need to complete the CPQ8-10. The instructions, as outlined on the front page of the questionnaire (see Appendix D and E), will be explained to the patients. They will be encouraged to reach out to the researcher (NFS) for clarification if any of the questions are unclear. This step will be repeated and patient has to fill in the same questionnaire every 3 months after treatment started.

   * T0 - before start treatment
   * 3 months after started treatment
   * 6 months after started treatment
   * 9 months after started treatment
5. Intervention 1 - PFM (protraction facemask) Patients assigned to intervention 1 will utilize the Petit protraction facemask from Dentamedik Sdn Bhd, in conjunction with a rapid maxillary expansion (RME). This facemask consists of a forehead pad and chin pad linked by a sturdy steel support rod. The RME will be affixed in the patient's mouth one week before activating the facemask, allowing the patient to adapt to the appliance. The design and components of the RME will adhere to standardized specifications An extraoral elastic band (Ormco Zoo Pack Elastics will be attached from the hook of the rapid maxillary expansion (RME) to the facemask rod, applying a forward force to the maxilla and ensuring the elastic crosses to prevent interference with the lips. The force vector is intended to pass through the maxilla center of resistance, and the point of force application should be distal to the lateral incisors, positioned in the canine-premolar area (Petit, 1983). The force position and direction should be inclined at an angle ranging from 20° to 30° to the occlusal plane (Petit, 1983). Patients will receive guidance to wear the Petit protraction facemask and elastics for 14-16 hours daily or as close to 24 hours as feasible (McNamara, 1987). The elastic force will be incrementally increased following the staggered approach proposed by Mandall in 2010.
6. Intervention 2 - UPFA

Upper partial fixed appliance / 2 by 4 appliance (refer figure 3.7) will be used in this study by using bracket set (119-142 Unitek™ Gemini Bracket MBT™ U/L 5x5 0T-Cuspid 3Hk) with molar bands (3M™ Victory Series™ First Molar Bands) or buccal tubes (3M™ Victory Series™ Superior Fit Buccal Tubes) and upper nickel titanium archwires (3M™ Unitek™ Nitinol Heat-activated Archwire) and upper stainless steel archwires (3M™ Unitek™ Permachrome Standard Archwire) . The archwire sequence are listed below:

1. 016 nickel titanium archwire

   • To start with 014 nickel titanium as first archwire in a severely rotated cases
2. 018 stainless steel archwire A metal/plastic tubing will be used to protect the soft nickel titanium archwire and a niti push coil will be used on stainless steel archwire to jump the bite. A bite riser will be cemented (self-cured Glass Ionomer Orthodontic cement, GC Fuji Ortho) on lower posterior teeth to disengage the occlusion to allow anterior crossbite correction.

7. Follow up review Patients will be reviewed every six weeks until anterior crossbite is corrected. Post-treatment records will be taken, and the appliance will be debonded. No retainers will be given as positive overjet with incisal overlap is considered stable.

ELIGIBILITY:
Inclusion Criteria:

1. Age group between 7 to 10 years
2. Three or four incisors in crossbite
3. Positive overbite
4. Class III skeletal with ANB equal to or less than 0 or retrusive maxilla
5. Amount of crowding equal to or less than 4 mm
6. Good oral hygiene

Exclusion Criteria:

1. Cleft lip and palate and/or craniofacial syndrome
2. Patients with syndromes or medical condition
3. Subjects involved in any other orthodontic trials
4. A maxilla-mandibular planes angle greater than 35 degree
5. Previous history of TMJ signs or symptoms
6. Lack of consent

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Skeletal changes | Before start treatment (issue appliance) and the end of treatment (after debond appliance) at 6 months to 9 months
  From Lateral cephalometric
  1. Skeletal changes in unit degree
  * SNA (°) - an increase at the end of treatment shows good treatment outcome
  * SNB (°) - no or minimal increase at the end of treatment shows good treatment outcome
  * ANB (°) - an increase at the end of treatment shows good treatment outcome
  * MMPA (°) - a minimal increase at the end of treatment is expected but not more than 35 degree shows a good treatment outcome
  * Upper incisor to maxillary plane angle (°) - an increase at the end of treatment shows good treatment outcome
  * Lower incisor to mandibular plane angle (°) - no changes or insignificant increase at the end of treatment shows good treatment outcome
  * Interincisal angle (°) - decrease at the end of treatment shows good treatment outcome
Skeletal changes | Before start treatment (issue appliance) and the end of treatment (after debond appliance) at 6 months to 9 months
  From lateral cephalometric
  - Increase or decrease in lower facial height (in percentage). Expected to have an increase after treatment but not more than 55 percent.
Dental changes | Before start treatment (issue appliance) and the end of treatment (after debond appliance) at 6 months to 9 months
  Study model to measure dental changes
  * Overjet (in milimeter) - an increase OJ at the end of treatment shows good treatment outcome
  * Overbite (in milimeter/ percentage) - a positive incisal overlap shows good treatment outcome for stability
Dental changes | Before start treatment (issue appliance) and the end of treatment (after debond appliance) at 6 months to 9 months
  Study model to measure canine and molar relationship changes based on British Standard Institution classification (Class I; Class II - 1/4 , 1/2, 3/4 , full ; Class III - 1/4 , 1/2, 3/4 , full)
  * Canine relationship - an improvement from Class III canine to Class I canine shows good treatment outcome
  * Molar relationship - an improvement from Class III molar to Class I molar shows good treatment outcome
Soft tissue changes | Before start treatment (issue appliance) and the end of treatment (after debond appliance) at 6 months to 9 months
  From lateral cephalometric
  • Nasolabial angle (°) - an improvement in naso labial angle near to 90 - 110 degree shows good treatment outcome
Soft tissue changes | Before start treatment (issue appliance) and the end of treatment (after debond appliance) at 6 months to 9 months
  From lateral cephalometric
  * Upper lip to E-line (in millimetres) - a decrease in millimetres to E-line shows good treatment outcome, less retrusive upper lips
  * Lower lip to E-line (in millimetres) - an improvement near to average value shows good treatment outcome (Milimetres can be increase or decrease depends on patients biting with mandibular displacement or not), averagely position lower lips

SECONDARY OUTCOMES:
Patients perception | From issuance appliance date to the end of treatment at 3 months, 6 months and after appliance removal
  Child Perception Questionnaire 8-10 will be used in this study to assess oral health-related quality of life scores for all participants at this time point:
  * before treatment,
  * 3 months after treatment
  * 6 months after treatment (if treatment not yet completed)
  * post- treatment A reduction/ decrease in the score at the end of treatment shows an improvement in oral health-related quality of life after the treatment is done.
Adverse effects | From issuance appliance date to the end of treatment at 3 months, 6 months and after appliance removal
  The number of breakages, injuries or any other adverse effects that happened throughout the treatment time will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Nur Farisya S Dr Nur Farisya Shamsuddin, Master in Oral Science, Principal Investigator — Faculty of Dentistry, Universiti Malaya
Locations (1):
- Faculty of Dentistry, Universiti Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
1. Protection of Patient Privacy: Ensuring the confidentiality of participants is a fundamental ethical obligation. Sharing identifiable information may risk the exposure of sensitive personal health data, which could lead to privacy breaches.
  2. Informed Consent Considerations: Participants in our study have provided informed consent with assurances that their personal and medical information will remain confidential and will not be shared beyond the scope of the study. Sharing identifiable patient data without explicit consent would violate this agreement.
  3. Minimizing Risks: Disclosing patient identification increases the potential risk of re-identification, even if other data elements are anonymized. To minimize any risk of harm to participants, we have opted not to share patient-specific identifiers.

REFERENCES:
- [Background] Mandall N, Cousley R, DiBiase A, Dyer F, Littlewood S, Mattick R, Nute SJ, Doherty B, Stivaros N, McDowall R, Shargill I, Worthington HV. Early class III protraction facemask treatment reduces the need for orthognathic surgery: a multi-centre, two-arm parallel randomized, controlled trial. J Orthod. 2016 Sep;43(3):164-75. doi: 10.1080/14653125.2016.1201302. PMID 27564126
- See also: A leaflet from British Orthodontic Society website — https://www.bos.org.uk/wp-content/uploads/2022/03/British-Orthodontic-Society-ProtractionHeadgearMarch2019.pdf